CLINICAL TRIAL: NCT02942654
Title: Pharmacokinetics and Glucodynamics of LY900014 Compared to Insulin Lispro Following Single-Dose Administration in Healthy Subjects
Brief Title: A Study of LY900014 Formulation in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 16170; I8B-MC-ITRL (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Results first posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2017-01

CONDITIONS: Healthy
MeSH Terms: interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY900014 (Experimental): Test formulation. 15-U dose of LY900014 administered subcutaneously (SC) in one of two periods.
  Interventions: Drug: LY900014
- Insulin Lispro (Active Comparator): Reference formulation. 15-U dose of Insulin Lispro administered SC in one of two periods.
  Interventions: Drug: Insulin Lispro

INTERVENTIONS:
Drug: LY900014 — Administered subcutaneously (SC)
  Other Names: Ultra-Rapid Lispro
  Arms: LY900014
Drug: Insulin Lispro — Administered SC
  Arms: Insulin Lispro

SUMMARY:
This study evaluates a new formulation of LY900014, a drug that lowers blood sugar. It is administered by injection under the skin of the abdomen. The study will be conducted in healthy people to investigate how quickly and how much LY900014 is absorbed and the effect of different doses of LY900014 on blood sugar levels. Side effects and tolerability will be documented. The study will last about 6 to 7 weeks for each participant, including screening and follow up. Screening is required within 28 days prior to entering the study.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy male or a female (not pregnant and agreeable to take birth control measures until study completion)
* Have a body mass index (BMI) of 18 to 30 kilogram per square meter (kg/m²), inclusive, at screening
* Have normal blood pressure, pulse rate, electrocardiogram (ECG), blood and urine laboratory test results that are acceptable for the study
* Are nonsmokers, have not smoked for at least 2 months prior to entering the study, and agree not to smoke (cigars, cigarettes, or pipes) or use smokeless tobacco for the duration of the study

Exclusion Criteria:

* Are currently participating in or completed a clinical trial within the last 30 days or any other type of medical research judged to be incompatible with this study
* Have previously participated or withdrawn from this study
* Have or used to have health problems or laboratory test results or ECG readings that, in the opinion of the doctor, could make it unsafe to participate, or could interfere with understanding the results of the study
* Had blood loss of more than 450 milliliters (mL) within the last month

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Singapore, Singapore

REFERENCES:
- [Derived] Leohr J, Dellva MA, Carter K, LaBell E, Linnebjerg H. Ultra Rapid Lispro (URLi) Accelerates Insulin Lispro Absorption and Insulin Action vs Humalog(R) Consistently Across Study Populations: A Pooled Analysis of Pharmacokinetic and Glucodynamic Data. Clin Pharmacokinet. 2021 Nov;60(11):1423-1434. doi: 10.1007/s40262-021-01030-0. Epub 2021 May 27. PMID 34041713

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of two treatment periods, with a minimum of 3 days washout period between each period.
Groups:
- Sequence 1: A single 15U dose of LY900014 or Insulin Lispro was administered subcutaneously (SC) as per the dosing schedule (Period 1: LY900014 ; Period 2: Insulin Lispro).
- Sequence 2: A single 15U dose of Insulin Lispro or LY900014 was administered subcutaneously (SC) as per the dosing schedule (Period 1: Insulin Lispro; Period 2: LY900014).
Period: Period 1
Arm/Group | Sequence 1 | Sequence 2
Started | 16 | 16
Received at Least 1 Dose of Study Drug | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0
Period: Washout
Arm/Group | Sequence 1 | Sequence 2
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Sequence 1 | Sequence 2
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Overall Study: Each participant was administered with 15 U dose of LY900014 and Insulin Lispro.
Arm/Group | Overall Study
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.0 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 32
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 32

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Insulin Lispro Area Under the Concentration Curve From Time Zero to 8 Hours (AUC[0-8 Hours])
Description: Area Under the Concentration Versus Time Curve (AUC) was measured from time zero to 8 hours (AUC[0-8 Hours]).
Time Frame: Predose (0), 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 55, 60, 70, 90, 120, 150, 180, 210, 240, 300, 330, 360, 420, and 480 minutes, post dose
Population: All randomized participants who receive at least 1 dose of study drug and have measurable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picomoles*hour/Liter (pmol*h/L)
Groups:
- LY900014: 15-U dose of LY900014 administered subcutaneously (SC) in one of two periods.
- Insulin Lispro: 15-U dose of Insulin Lispro administered SC in one of two periods.
Arm/Group | LY900014 | Insulin Lispro
Number analyzed (Participants) | 31 | 32
Picomoles*hour/Liter (pmol*h/L) | 2050 (18) | 1930 (19)

2. Secondary Outcome: Glucodynamics (GD): Total Amount of Glucose Infused (Gtot)
Description: Gtot is used to measure the study drug action over time as measured by the euglycaemic clamp procedure. During the euglycaemic clamp procedure, blood glucose concentrations are held constant after the administration of LY900014 or Insulin Lispro by adjusting the exogenous glucose infusion rate. Data presented were adjusted by the body weight.
Time Frame: 2.5 minutes for the first 30 minutes, then every 5 minutes until 120 minutes postdose, and then every 10 minutes until 480 minutes postdose
Population: All randomized participants who received at least one dose of study drug and have evaluable glucodynamic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligrams (mg)
Arm/Group | LY900014 | Insulin Lispro
Number analyzed (Participants) | 32 | 32
Milligrams (mg) | 115000 (32) | 125000 (34)

ADVERSE EVENTS:
Description: All randomized participants who received at least one dose of the study drug.
Arm/Group | LY900014 | Insulin Lispro
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 3/32 | 7/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY900014 (N=32) | Insulin Lispro (N=32)
Catheter site bruise (General disorders) | 0 (0) | 2 (2)
Infusion site bruising (General disorders) | 1 (1) | 2 (2)
Injection site erythema (General disorders) | 2 (2) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 2 (2)
Vessel puncture site swelling (General disorders) | 0 (0) | 2 (3)
Headache (Nervous system disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes